CLINICAL TRIAL: NCT06455345
Title: Advancing Online Psychology Tools for the Transitional Pain Service (ADOPT-TPS): Pilot Feasibility and Efficacy Randomized-Controlled Trial of a Scalable, Online Psychology Intervention for Post-Surgical Pain and Opioid Use
Brief Title: Online Psychology Program for Chronic Pain After Surgery
Acronym: ADOPT-TPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other); York University (Other); Toronto General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-5934; MSU-23-002 (Other Grant/Funding Number: Academic Health Sciences Centre - Innovation Fund)
Record Dates: First submitted 2023-12-27; First posted 2024-06-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Post-surgical Pain; Pain, Acute; Pain, Chronic; Post-Surgical Pain, Chronic
Keywords: Feasibility Studies; Digital Health; Acceptance and Commitment Therapy; Mindfulness; Internet-based Intervention; Randomized Controlled Trial
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The present study will evaluate whether the self-guided online ADOPT-TPS tool is a the feasible and efficacious intervention compared to the psychologist-guided group workshop.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Only the participants and the research coordinator will know which group (self-guided vs. psychologist-guided) an individual participant will be randomly assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-guided Online ACT (Experimental): The intervention is a self-guided ACT program delivered on an online platform. The program is developed based on the psychologist-guided ACT group intervention for chronic pain and opioid use after surgery.
  Interventions: Device: Self-Guided Online ACT Program
- Psychologist-guided Online ACT (Active Comparator): The psychologist-guided ACT group workshop is an evidence-based psychology intervention for chronic pain and opioid use after surgery.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Device: Self-Guided Online ACT Program — Participants will be invited to access the ACT program on the Manage My Pain (MMP) app. Participants will follow the instructions in the app to complete the program in a self-paced manner. The program includes psychoeducational materials, guided mindfulness meditations, and self-reflection activities.
  Arms: Self-guided Online ACT
Other: Treatment As Usual — Participants will be invited to join a one-session ACT group workshop guided by a psychologist. The session will take place virtually using video call software. The psychologist will guide participants through the workshop agenda, which will include psychoeducational material, guided mindfulness meditations, and partaking in voluntary discussions with other group members.
  Other Names: Psychologist-guided online ACT
  Arms: Psychologist-guided Online ACT

SUMMARY:
This project will evaluate the feasibility of a new fully self-guided online Acceptance and Commitment Therapy (ACT) program entitled Advancing Online Psychology Tools for the Transitional Pain Service (ADOPT-TPS), developed on an online health application platform called Manage My Pain (MMP). The ACT program is designed to teach mindfulness skills and provide psychoeducation about post-surgical pain. The feasibility of the self-guided online program will be compared to a pre-existing psychologist-guided workshop that delivers the same program. It is anticipated that the self-guided online ACT program will be deemed feasible by participants.

DETAILED DESCRIPTION:
The Transitional Pain Service (TPS) at Toronto General Hospital is a multidisciplinary treatment program that aims to prevent chronic post-surgical pain (CPSP) and persistent opioid use after surgery. CPSP is a major public health concern impacting from 10% up to 70% of patients, depending on the type of surgery. Those experiencing CPSP are at higher risk for prolonged opioid use, which introduces challenges like addiction, misuse, and overdose. Acceptance and Commitment Therapy (ACT) is an evidence-based psychology intervention that is effective in reducing patients' risk of CPSP and opioid use. However, access to this intervention is currently limited to predominantly in-person, specialized hospital-based clinic settings like the TPS, which prioritize patients at highest risk for CPSP and often require physician referrals for quick access. There is a need for such treatment approaches to spread to other institutions and to be available for lower-risk post-surgery patients, yet the shortage of specialized pain psychologists creates a barrier to widespread dissemination. The current project will evaluate the feasibility of a novel fully self-guided online ACT intervention entitled Advancing Online Psychology Tools for the Transitional Pain Service (ADOPT-TPS), developed on a mobile health application platform called Manage My Pain (MMP). A randomized, controlled pilot feasibility trial will evaluate the efficacy of ADOPT-TPS by comparing it to a pre-existing psychologist-guided workshop. Once tested, this scalable, evidence-based online intervention can be easily implemented at institutions across Canada and beyond to address CPSP and opioid use without the need for specialized pain psychologists on staff.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a post-surgical referral to the TPS
* Patients who have access to a device that can connect to the Internet

Exclusion Criteria:

* Patients who have received TPS psychology treatment
* Patients with a known history of serious mental illness (e.g., psychosis and/or active mania)
* Patients who have limited comprehension of English or comprehension deficits due to dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the online ACT program as assessed by the Feasibility Survey | Participants will be sent a link to fill out the measure within 1 week of completing their respective program.
  A 10-item Likert scale (min possible score = 10, max possible score = 70). Higher scores indicate greater feasibility.
Acceptability of the online ACT program as assessed by the Treatment Evaluation Inventory - Short Form | Participants will be sent a link to fill out the measure within 1 week of completing their respective program.
  A 9-item Likert scale (min possible score = 9, max possible score = 45). Higher scores indicate greater acceptability.
Retrospective Semi-structured Interview | Participants will be sent an invitation for an interview within 1 month after completing their respective program
  A brief interview with a randomized subset of participants
Treatment Adherence as assessed by the Integration of ACT Skills Survey | Participants will be sent a link to complete the measure within 1 month after completing their respective program.
  A 5-item Likert scale (min possible score = 5, max possible score = 35). Higher scores indicate greater treatment adherence

SECONDARY OUTCOMES:
Pain Intensity as assessed by the Pain Numerical Rating Scale | Participants will be sent a link to fill out the measure prior to starting their respective program, within 1 week of completing their respective program, and 1 month after completing their respective program.
  A 4-item Likert scale (min possible score = 0, max possible score = 40). Higher scores indicate greater pain intensity.
Pain Interference as assessed by the PROMIS Pain Interference Scale - Short Form 8a | Participants will be sent a link to fill out the measure prior to starting their respective program, within 1 week of completing their respective program, and 1 month after completing their respective program.
  A 8-item Likert scale (min possible score = 8, max possible score = 40). Higher scores indicate greater pain interference.
Pain Medication Misuse as assessed by the PROMIS Prescription Pain Medication Misuse Scale - Short Form 7a | Participants will be sent a link to fill out the measure prior to starting their respective program, within 1 week of completing their respective program, and 1 month after completing their respective program.
  A 7-item Likert scale (min possible score = 7, max possible score = 5). Higher scores indicate greater pain medication misuse.
Pain Catastrophizing as assessed by the Pain Catastrophizing Scale | Participants will be sent a link to fill out the measure prior to starting their respective program, within 1 week of completing their respective program, and 1 month after completing their respective program.
  A 13-item Likert scale (min possible score = 0, max possible score = 52). Higher scores indicate greater pain catastrophizing.
Depressive symptoms as assessed by PROMIS Emotional Distress - Depression - Short Form 8b | Participants will be sent a link to fill out the measure prior to starting their respective program, within 1 week of completing their respective program, and 1 month after completing their respective program.
  A 8-item Likert scale (min possible score = 8, max possible score = 40). Higher scores indicate greater depressive symptoms.
Anxiety symptoms as assessed by the PROMIS Emotional Distress - Anxiety - Short Form 8A | Participants will be sent a link to fill out the measure prior to starting their respective program, within 1 week of completing their respective program, and 1 month after completing their respective program.
  A 8-item Likert scale (min possible score = 8, max possible score = 40). Higher scores indicate greater anxiety symptoms.
Psychological Inflexibility in Pain as measured by the Psychological Inflexibility in Pain Scale | Participants will be sent a link to fill out the measure prior to starting their respective program, within 1 week of completing their respective program, and 1 month after completing their respective program.
  A 16-item Likert scale (min possible score = 16, max possible score = 112). Higher scores indicate greater psychological inflexibility in pain.
Use of Study Platform as assessed by the Use of Manage My Pain Platform Survey | Participants will be sent a link to fill out the measure within 1 week of completing the respective program, and 1 month after completing their respective program.
  A 5-item Likert scale (min possible score = 4, max possible score = 20). Higher scores indicate more frequent use of the platform.

CONTACTS AND LOCATIONS:
Overall Officials: Maxwell Slepian, PhD, C Psych, Principal Investigator — Toronto General Hospital
Locations (2):
- Canada (2):
  - Toronto General Hospital- The Department of Anesthesia and Pain Management, Toronto, Ontario
  - University Health Network- Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Relevant de-identified study data will be shared upon request.
Time Frame: The data will become available after primary outcomes manuscript is published and will remain available for 10 years.
Access Criteria: Request for access will be reviewed by the principle investigator and the study team and will be granted in accordance with University Health Network policies.

REFERENCES:
- [Background] Katz J, Weinrib A, Fashler SR, Katznelzon R, Shah BR, Ladak SS, Jiang J, Li Q, McMillan K, Santa Mina D, Wentlandt K, McRae K, Tamir D, Lyn S, de Perrot M, Rao V, Grant D, Roche-Nagle G, Cleary SP, Hofer SO, Gilbert R, Wijeysundera D, Ritvo P, Janmohamed T, O'Leary G, Clarke H. The Toronto General Hospital Transitional Pain Service: development and implementation of a multidisciplinary program to prevent chronic postsurgical pain. J Pain Res. 2015 Oct 12;8:695-702. doi: 10.2147/JPR.S91924. eCollection 2015. PMID 26508886
- [Background] Fletcher D, Stamer UM, Pogatzki-Zahn E, Zaslansky R, Tanase NV, Perruchoud C, Kranke P, Komann M, Lehman T, Meissner W; euCPSP group for the Clinical Trial Network group of the European Society of Anaesthesiology. Chronic postsurgical pain in Europe: An observational study. Eur J Anaesthesiol. 2015 Oct;32(10):725-34. doi: 10.1097/EJA.0000000000000319. PMID 26241763
- [Background] Schug SA, Lavand'homme P, Barke A, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic postsurgical or posttraumatic pain. Pain. 2019 Jan;160(1):45-52. doi: 10.1097/j.pain.0000000000001413. PMID 30586070
- [Background] Rosenberger DC, Pogatzki-Zahn EM. Chronic post-surgical pain - update on incidence, risk factors and preventive treatment options. BJA Educ. 2022 May;22(5):190-196. doi: 10.1016/j.bjae.2021.11.008. Epub 2022 Feb 24. No abstract available. PMID 35496645
- [Background] Katz J, Weinrib AZ, Clarke H. Chronic postsurgical pain: From risk factor identification to multidisciplinary management at the Toronto General Hospital Transitional Pain Service. Can J Pain. 2019 Jul 30;3(2):49-58. doi: 10.1080/24740527.2019.1574537. eCollection 2019. PMID 35005419
- [Background] Clarke H, Soneji N, Ko DT, Yun L, Wijeysundera DN. Rates and risk factors for prolonged opioid use after major surgery: population based cohort study. BMJ. 2014 Feb 11;348:g1251. doi: 10.1136/bmj.g1251. PMID 24519537
- [Background] Clarke H, Azargive S, Montbriand J, Nicholls J, Sutherland A, Valeeva L, Boulis S, McMillan K, Ladak SSJ, Ladha K, Katznelson R, McRae K, Tamir D, Lyn S, Huang A, Weinrib A, Katz J. Opioid weaning and pain management in postsurgical patients at the Toronto General Hospital Transitional Pain Service. Can J Pain. 2018 Aug 20;2(1):236-247. doi: 10.1080/24740527.2018.1501669. eCollection 2018. PMID 35005382
- [Background] Abid Azam M, Weinrib AZ, Montbriand J, Burns LC, McMillan K, Clarke H, Katz J. Acceptance and Commitment Therapy to manage pain and opioid use after major surgery: Preliminary outcomes from the Toronto General Hospital Transitional Pain Service. Can J Pain. 2017 Jun 28;1(1):37-49. doi: 10.1080/24740527.2017.1325317. eCollection 2017. PMID 35005340
- [Background] Dindo L, Zimmerman MB, Hadlandsmyth K, StMarie B, Embree J, Marchman J, Tripp-Reimer T, Rakel B. Acceptance and Commitment Therapy for Prevention of Chronic Postsurgical Pain and Opioid Use in At-Risk Veterans: A Pilot Randomized Controlled Study. J Pain. 2018 Oct;19(10):1211-1221. doi: 10.1016/j.jpain.2018.04.016. Epub 2018 May 17. PMID 29777950
- [Background] Buhrman M, Skoglund A, Husell J, Bergstrom K, Gordh T, Hursti T, Bendelin N, Furmark T, Andersson G. Guided internet-delivered acceptance and commitment therapy for chronic pain patients: a randomized controlled trial. Behav Res Ther. 2013 Jun;51(6):307-15. doi: 10.1016/j.brat.2013.02.010. Epub 2013 Mar 14. PMID 23548250
- [Background] Scott W, Chilcot J, Guildford B, Daly-Eichenhardt A, McCracken LM. Feasibility randomized-controlled trial of online Acceptance and Commitment Therapy for patients with complex chronic pain in the United Kingdom. Eur J Pain. 2018 Apr 28. doi: 10.1002/ejp.1236. Online ahead of print. PMID 29704880
- [Background] Hayes S, Hogan M, Dowd H, Doherty E, O'Higgins S, Nic Gabhainn S, MacNeela P, Murphy AW, Kropmans T, O'Neill C, Newell J, McGuire BE. Comparing the clinical-effectiveness and cost-effectiveness of an internet-delivered Acceptance and Commitment Therapy (ACT) intervention with a waiting list control among adults with chronic pain: study protocol for a randomised controlled trial. BMJ Open. 2014 Jul 2;4(7):e005092. doi: 10.1136/bmjopen-2014-005092. PMID 24993763
- [Background] Trindade IA, Guiomar R, Carvalho SA, Duarte J, Lapa T, Menezes P, Nogueira MR, Patrao B, Pinto-Gouveia J, Castilho P. Efficacy of Online-Based Acceptance and Commitment Therapy for Chronic Pain: A Systematic Review and Meta-Analysis. J Pain. 2021 Nov;22(11):1328-1342. doi: 10.1016/j.jpain.2021.04.003. Epub 2021 Apr 20. PMID 33892153
- [Background] Cuijpers P, van Straten A, Andersson G. Internet-administered cognitive behavior therapy for health problems: a systematic review. J Behav Med. 2008 Apr;31(2):169-77. doi: 10.1007/s10865-007-9144-1. PMID 18165893
- [Background] Fox MP. A systematic review of the literature reporting on studies that examined the impact of interactive, computer-based patient education programs. Patient Educ Couns. 2009 Oct;77(1):6-13. doi: 10.1016/j.pec.2009.02.011. Epub 2009 Apr 3. PMID 19345550
- [Background] Lin J, Klatt LI, McCracken LM, Baumeister H. Psychological flexibility mediates the effect of an online-based acceptance and commitment therapy for chronic pain: an investigation of change processes. Pain. 2018 Apr;159(4):663-672. doi: 10.1097/j.pain.0000000000001134. PMID 29320375
- [Background] Simister HD, Tkachuk GA, Shay BL, Vincent N, Pear JJ, Skrabek RQ. Randomized Controlled Trial of Online Acceptance and Commitment Therapy for Fibromyalgia. J Pain. 2018 Jul;19(7):741-753. doi: 10.1016/j.jpain.2018.02.004. Epub 2018 Mar 2. PMID 29481976
- [Background] Lin J, Scott W, Carpenter L, Norton S, Domhardt M, Baumeister H, McCracken LM. Acceptance and commitment therapy for chronic pain: protocol of a systematic review and individual participant data meta-analysis. Syst Rev. 2019 Jun 14;8(1):140. doi: 10.1186/s13643-019-1044-2. PMID 31200768
- [Background] van de Graaf DL, Trompetter HR, Smeets T, Mols F. Online Acceptance and Commitment Therapy (ACT) interventions for chronic pain: A systematic literature review. Internet Interv. 2021 Oct 1;26:100465. doi: 10.1016/j.invent.2021.100465. eCollection 2021 Dec. PMID 34660209
- [Background] Veehof MM, Oskam MJ, Schreurs KMG, Bohlmeijer ET. Acceptance-based interventions for the treatment of chronic pain: a systematic review and meta-analysis. Pain. 2011 Mar;152(3):533-542. doi: 10.1016/j.pain.2010.11.002. Epub 2011 Jan 19. PMID 21251756
- [Background] Weinrib A, Azam MA, Latman VV, Janmohamed T, Clarke H, Katz J. Manage My Pain: A Patient-Driven Mobile Platform to Prevent and Manage Chronic Postsurgical Pain. Novel Applications of Virtual Communities in Healthcare Settings. doi:10.4018/978-1-5225-2958-3.ch004
- [Background] Slepian PM, Peng M, Janmohamed T, Kotteeswaran Y, Manoo V, Blades AM, Fiorellino J, Katznelson R, Tamir D, McRae K, Kahn M, Huang A, Kona S, Thaker S, Weinrib A, Katz J, Clarke H. Engagement with Manage My Pain mobile health application among patients at the Transitional Pain Service. Digit Health. 2020 Oct 13;6:2055207620962297. doi: 10.1177/2055207620962297. eCollection 2020 Jan-Dec. PMID 33117557
- See also: The home webpage for ManagingLife, the company that will host the ACT For My Pain intervention on the digital application (Manage My Pain). — https://managinglife.com